CLINICAL TRIAL: NCT02784054
Title: Reduced-dose Radiotherapy Following High-dose Chemotherapy and Autologous Stem Cell Transplantation in Patients With Central Nervous System Non-germinomatous Germ Cell Tumors
Brief Title: Reduced Dose Radiotherapy Following High Dose Chemotherapy in Intracranial Non-germinomatous Germ Cell Tumor
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-07-146
Record Dates: First submitted 2016-05-24; First posted 2016-05-26 (Estimated); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Intracranial Non-germinomatous Germ Cell Tumor
MeSH Terms: interventions — Carboplatin; Etoposide; Cyclophosphamide; Bleomycin; Thiotepa; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intracranial NGGCT (Experimental): 1. Six cycles of chemotherapy with carboplatin, etoposide, bleomycin (CEB) and cyclophosphamide, etoposide, bleomycin (CyEB) regimen.
  2. Peripheral blood stem cell collection during the first cycle of chemotherapy.
  3. Surgery, if there is residual tumor after chemotherapy.
  4. Tandem high dose chemotherapy (HDCT) and autologous stem cell transplantation (auto-SCT)
     * 1st HDCT: Carboplatin, thiotepa, etoposide
     * 2nd HDCT: Cyclophosphamide, melphalan
  5. Reduced dose of radiotherapy
  Interventions: Drug: Carboplatin; Drug: Etoposide; Drug: Cyclophosphamide; Drug: Bleomycin; Drug: Thiotepa; Drug: Melphalan; Radiation: Reduced dose radiotherapy

INTERVENTIONS:
Drug: Carboplatin
Drug: Etoposide
Drug: Cyclophosphamide
Drug: Bleomycin
Drug: Thiotepa
Drug: Melphalan
Radiation: Reduced dose radiotherapy

SUMMARY:
The purpose of this study is to evaluate the outcome of intracranial non-germinomatous germ cell tumor (NGGCT) treated with reduced radiotherapy following high dose chemotherapy and autologous stem cell transplantation (HDCT/auto-SCT).

DETAILED DESCRIPTION:
Treatment outcome of intracranial NGGCT is around 50% with conventional chemo- and radiotherapy. Also, late sequelae such as endocrinopathy or cognitive problem are unavoidable especially with craniospinal irradiation. In this study, high dose chemotherapy and reduced dose of radiotherapy will be used to improve survival and minimize the late sequelae in the patients with intracranial NGGCT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically proven intracranial non-germinomatous germ cell tumor or
* Patients who have brain mass which are suspected as intracranial germ cell tumor and elevated serum or cerebrospinal fluid alpha-feto protein.

Exclusion Criteria:

* Patients with organ dysfunction (ejection fraction <40%, creatinine > 3 x upper limit of normal (ULN), aspartate aminotransferase/alanine aminotransaminase > 5 x ULN).
* Pregnant or nursing women

Ages: 3 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2014-04; Primary Completion 2021-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Rate of event free survival | Up to 3 years

SECONDARY OUTCOMES:
Rate of late adverse events | Up to 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea